CLINICAL TRIAL: NCT06893133
Title: Personalized ctDNA-MRD in Recurrence Monitoring for Gastric Cancer Patients Undergoing Perioperative Treatment Combined With Curative Surgical Resection
Brief Title: ctDNA-MRD Monitoring After Resection in Gastric Cancer
Acronym: MRD-GC
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Chief Physician, Peking University Cancer Hospital & Institute
Other Study IDs: 2025KT40
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
Keywords: ctDNA; MRD; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Preoperative drug therapy combined with R0 resection in patients with gastric cancer: Names: MRD testing Description: MRD refers to the small, residual number of cancer cells that remain in a patient's body after treatment, often undetectable by conventional methods, but detectable using ctDNA. MRD-positive indicates the presence of residual disease, while MRD-negative suggests potential cure.

SUMMARY:
Numerous studies have demonstrated that circulating tumor DNA (ctDNA)-based molecular residual disease (MRD) detection has significant clinical value in postoperative recurrence monitoring, adjuvant treatment decision-making, and early intervention. Our previous retrospective study, using fixed ctDNA-MRD, confirmed that postoperative ctDNA-MRD can predict recurrence risk. Therefore, we plan to conduct a further prospective, multicenter, observational study, utilizing a combination of personalized ctDNA-MRD and fixed MRD panels, to dynamically monitor gastric cancer patients who have received neoadjuvant therapy followed by curative resection. The study will systematically analyze the correlation between ctDNA-MRD status and tumor recurrence and metastasis, assess its sensitivity and specificity in recurrence prediction, and compare its early warning advantage over traditional imaging techniques in predicting recurrence.

DETAILED DESCRIPTION:
China has the highest incidence and mortality rates of gastric cancer in the world, with approximately 70% of patients diagnosed at an advanced stage. Perioperative treatment combined with surgery is the recommended treatment approach for advanced gastric cancer. However, a considerable proportion of patients still experience recurrence and metastasis after surgery. Imaging studies are the standard method for monitoring postoperative recurrence and metastasis, but they can only detect recurrence once the metastatic lesions have grown to a certain size. In contrast, ctDNA-MRD testing can detect residual tumor molecular signals in the blood, providing early signs of recurrence and allowing for timely intervention while the tumor is still in its "incipient stage." Previous clinical data have shown that MRD testing can identify recurrent and metastatic patients months earlier than traditional imaging methods, with the median lead time varying by cancer type: 9.5 months for breast cancer, 8.7 months for colon cancer, 5.2 months for lung cancer, and 2.8 months for bladder cancer.

Therefore, we plan to conduct a further prospective, multicenter, observational study, utilizing a combination of personalized ctDNA-MRD and fixed MRD panels, to dynamically monitor gastric cancer patients who have received neoadjuvant therapy followed by curative resection. The study will systematically analyze the correlation between ctDNA-MRD status and tumor recurrence and metastasis, assess its sensitivity and specificity in recurrence prediction, and compare its early warning advantage over traditional imaging techniques in predicting recurrence. In addition, this project will focus on establishing and improving a dynamic MRD monitoring system, laying the foundation for future interventional clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have received neoadjuvant therapy and radical resection (R0).
2. Pathologically confirmed ypTNM stage II-III gastric or gastroesophageal junction adenocarcinoma.
3. Patients must be able to provide sufficient fresh tissue/biopsies or minimum 5-10 FFPE sections for NGS-WES analysis.
4. Patients must be able to follow the study visit schedule and be willing to cooperate with the study by providing blood samples at the indicated time point.

Exclusion Criteria:

1. Patients who could not receive enhanced CT, gastroscopy and other routine review after surgery.
2. Patients who could not perform WES or ctDNA-MRD detection for various reasons after surgery.
3. Other cases considered unsuitable for inclusion by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 110 patients with gastric cancer undergoing preoperative drug therapy combined with R0 resection were enrolled.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Predictive Accuracy of Personalized ctDNA-MRD for Postoperative Recurrence | From the time of surgical resection to the point of resurrence within 2 years
  Sensitivity, Specificity, and Positive predictive value of ctDNA-MRD in predicting postoperative recurrence

SECONDARY OUTCOMES:
Lead time of personalized ctDNA-MRD compared to radiologic surveillance in postoperative recurrence prediction | From ctDNA-MRD positive to the point of CT imaging showing recurrence
  Time interval between ctDNA-MRD positivity and imaging diagnosis of recurrence

OTHER OUTCOMES:
Prognostic or recurrence molecular biomarkers | From the time of surgical resection to the point of recurrence within 2 years
  Prognostic or recurrence molecular biomarkers associated with postoperative recurrence and metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Tarazona N, Gimeno-Valiente F, Gambardella V, Zuniga S, Rentero-Garrido P, Huerta M, Rosello S, Martinez-Ciarpaglini C, Carbonell-Asins JA, Carrasco F, Ferrer-Martinez A, Bruixola G, Fleitas T, Martin J, Tebar-Martinez R, Moro D, Castillo J, Espi A, Roda D, Cervantes A. Targeted next-generation sequencing of circulating-tumor DNA for tracking minimal residual disease in localized colon cancer. Ann Oncol. 2019 Nov 1;30(11):1804-1812. doi: 10.1093/annonc/mdz390. PMID 31562764
- [Background] Christensen E, Birkenkamp-Demtroder K, Sethi H, Shchegrova S, Salari R, Nordentoft I, Wu HT, Knudsen M, Lamy P, Lindskrog SV, Taber A, Balcioglu M, Vang S, Assaf Z, Sharma S, Tin AS, Srinivasan R, Hafez D, Reinert T, Navarro S, Olson A, Ram R, Dashner S, Rabinowitz M, Billings P, Sigurjonsson S, Andersen CL, Swenerton R, Aleshin A, Zimmermann B, Agerbaek M, Lin CJ, Jensen JB, Dyrskjot L. Early Detection of Metastatic Relapse and Monitoring of Therapeutic Efficacy by Ultra-Deep Sequencing of Plasma Cell-Free DNA in Patients With Urothelial Bladder Carcinoma. J Clin Oncol. 2019 Jun 20;37(18):1547-1557. doi: 10.1200/JCO.18.02052. Epub 2019 May 6. PMID 31059311
- [Background] Chaudhuri AA, Chabon JJ, Lovejoy AF, Newman AM, Stehr H, Azad TD, Khodadoust MS, Esfahani MS, Liu CL, Zhou L, Scherer F, Kurtz DM, Say C, Carter JN, Merriott DJ, Dudley JC, Binkley MS, Modlin L, Padda SK, Gensheimer MF, West RB, Shrager JB, Neal JW, Wakelee HA, Loo BW Jr, Alizadeh AA, Diehn M. Early Detection of Molecular Residual Disease in Localized Lung Cancer by Circulating Tumor DNA Profiling. Cancer Discov. 2017 Dec;7(12):1394-1403. doi: 10.1158/2159-8290.CD-17-0716. Epub 2017 Sep 24. PMID 28899864
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300